CLINICAL TRIAL: NCT01483092
Title: Inulin Modifies Gut Microbiota, Fecal Lactate Concentration and Fecal pH But Does Not Influence Iron Absorption in Women With Low Iron Status
Brief Title: Effect of Inulin on Iron Absorption in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Prof., Swiss Federal Institute of Technology
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: INOL
Record Dates: First submitted 2011-11-09; First posted 2011-12-01 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-06

CONDITIONS: Iron Absorption; Gut Bacteria
MeSH Terms: interventions — Inulin; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- inulin (Experimental)
  Interventions: Dietary Supplement: inulin
- maltodextrin (Placebo Comparator)
  Interventions: Dietary Supplement: maltodextrin

INTERVENTIONS:
Dietary Supplement: inulin — 20g/day for 4 weeks
  Arms: inulin
Dietary Supplement: maltodextrin — 20g/day for 4 weeks
  Arms: maltodextrin

SUMMARY:
Prebiotics are non-digestible food ingredients that beneficially affect the host by selectively stimulating the growth or activity of species in the colon that can improve host health.

Inulin-type fructans (inulin and oligofructose) are natural food ingredients with prebiotic activity. Fermentation of inulin and oligofructose by lactic acid producing bacteria results in an increase in bacterial biomass and the production of SCFA (acetate, propionate and butyrate), lactic acid and the gases CO2 and H2. They are naturally present in significant amounts in several vegetables such as garlic, artichoke, onion, asparagus, leek and wheat (1-4%). Based on consumption data, the daily intake of inulin in Europe varies between 3.2 and 11.3g mainly from wheat (2-7.8g/d). However, this might have changed recently since inulin and oligofructose are used by the food industry either as sucrose and fat replacements or due to their health benefits for the human host.

Several human absorption studies evaluated the effect of inulin/oligofructose on mineral absorption. It was shown that calcium and magnesium absorption was positively influenced. Until now, the positive effect on iron absorption was only shown in animals. The influence on human iron absorption was investigated twice. Both studies reported no effect of inulin/oligofructose on iron absorption, but this was most likely due to poorly conceived study designs.

The aim of the present study is to demonstrate that inulin consumption over several weeks can lead to enhanced iron absorption in humans under optimized conditions.

ELIGIBILITY:
Inclusion Criteria:

* non-pregnant, non-lactating women
* between 18 and 40 years
* below 65kg

Exclusion Criteria:

* metabolic, chronic and gastro-intestinal disease
* long-term medication
* blood donation within 6 month before the study-

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2011-08; Primary Completion 2011-11 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
impact of inulin on iron absorption from standardized test meals, measured in humans by stable iron isotope technique | 3 month

SECONDARY OUTCOMES:
impact of inulin on the concentration of gut microbiota (bifidobacteria and total bacteria), SCFA and fecal pH in human subjects | 3 month
  Concentration of bifidobacteria, total bacteria, SCFA (acetate, propionate, butyrate, formate), lactate, and pH will be measured (in the fecal samples of study participants) and compared between baseline, inulin period and placebo period. The pH of fecal sqamples will be measured using a digital pH meter. HPLC measurements will be done for the determination of SCFA and lactate. DNA amplification and detection will be done by quantitative PCR.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Hurrell, Prof. Dr., Principal Investigator — ETH Zurich
Locations (1):
- ETH, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Petry N, Egli I, Chassard C, Lacroix C, Hurrell R. Inulin modifies the bifidobacteria population, fecal lactate concentration, and fecal pH but does not influence iron absorption in women with low iron status. Am J Clin Nutr. 2012 Aug;96(2):325-31. doi: 10.3945/ajcn.112.035717. Epub 2012 Jun 27. PMID 22743314